CLINICAL TRIAL: NCT01387334
Title: The Effectiveness of a Home-Based Resistance Exercise Training Program With Rubber Bands for Glycemic Control in Individuals With Type 2 Diabetes Mellitus
Brief Title: The Effectiveness of Resistance Exercise for Glycemic Control in Type 2 Diabetes Mellitus Patients
Acronym: RE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Department of Community Medicine, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prince of Songkla University
Record Dates: First submitted 2011-06-13; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes
Keywords: resistive exercise; Resistance Exercise Training Program; Rubber Bands; Glycemic Control; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resistance Exercise Training Program (Experimental)
  Interventions: Behavioral: Resistance Exercise Training Program With Rubber Bands

INTERVENTIONS:
Behavioral: Resistance Exercise Training Program With Rubber Bands — Resistive exercise consist of 5-min warm up, at least 30 min resistive exercise using rubber band as recommendation (8-12 times per set, at least 3 sets per day and at least 3 days per week) and 5-min cool down
  Other Names: elastic band

SUMMARY:
Resistance exercise is effective in improving glycemic control in diabetes patients. The effectiveness of a home-based resistance exercise program has not been establish.

DETAILED DESCRIPTION:
Exercise play an important role in diabetes control. The American Diabetes Association (ADA) approved of resistive exercise as an effective method in controlling blood sugar of type 2 diabetes patients. Few community-based intervention has been establish. So the authors developed the low-cost community based resistance exercise program to promote exercise in of type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes was diagnosed by physician using fasting plasma glucose not less than 126 mg/dl and/or HbA1c not less than 7 %.
* Type 2 diabetes was diagnosed at least 6 months previously.
* The subject was ongoing treatment in primary care unit of prince of Songkla University.

Exclusion Criteria:

* Gestational diabetes and type 1 diabetes patients
* History of cardiovascular disease within the pass 6 months or any unstable chronic condition including dementia, proliferative diabetic retinopathy, retinal hemorrhage or detachment, dialysis and diabetic foot patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
compliance of home-based resistive exercise training | 3 years
  The home visit and telephone call was done to follow up the compliance of home-based resistive exercise training during 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Thanitha Sirirak, MD, Principal Investigator — Department of Community Medicine, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand